CLINICAL TRIAL: NCT05188365
Title: Acupuncture Efficacy on Lipids in Tinnitus Patients With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003525
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Tinnitus, Subjective; Obesity; Lipids
MeSH Terms: conditions — Tinnitus; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): different body acupuncture points will be selected to be manually punctured in addition to 4 acupoints on the skin of abdominal surface (the four points will be electrical stimulated during acupuncture). the session (20 minutes) will repeated thrice weekly. the total duration of the study will be 60 days.
  The points that will be manually acupunctured all over the body of every patient will be: SJ(3)/SJ(5)/SJ(17)/SJ(18)/SJ(19)/SJ(20)/SJ(21)/SJ(22)/GB(2)/GB(8)/GB(20)/LI(4)/LI(11)/KI(3)/SP(6)/ST(36)/REN(4)/REN(9)/REN(12)
  The acupuncture points that will be electrically stimulated on the abdomen of every patient will be: bilateral Stomach 25 in addition to gallbladder 28 acupoints.
  Interventions: Other: true acupuncture
- Group B (Sham Comparator): different body acupuncture points will be selected to be manually punctured in addition to 4 acupoints on the skin of abdominal surface (the four points will be electrical stimulated during acupuncture). opposite to group A, in this group, the acupuncture needles will be inserted manually and very adjacent to the real location of group-A acupoints (sham acupuncture). The electrical stimulator will connected to abdominal acupoints (bilateral Stomach 25 in addition to gallbladder 28 acupoints) but it will be turned off during the sessions. the session will repeated thrice weekly. the total duration of the study will be 60 days.
  Interventions: Other: sham acupuncture

INTERVENTIONS:
Other: true acupuncture — different body acupuncture points will be selected to be manually punctured in addition to 4 acupoints on the skin of abdominal surface (the four points will be electrical stimulated during acupuncture). the session (20 minutes) will repeated thrice weekly. the total duration of the study will be 60 days.
  The points that will be manually acupunctured all over the body of every patient will be: SJ(3)/SJ(5)/SJ(17)/SJ(18)/SJ(19)/SJ(20)/SJ(21)/SJ(22)/GB(2)/GB(8)/GB(20)/LI(4)/LI(11)/KI(3)/SP(6)/ST(36)/REN(4)/REN(9)/REN(12)
  The acupuncture points that will be electrically stimulated on the abdomen of every patient will be: bilateral Stomach 25 in addition to gallbladder 28 acupoints.
  Arms: group A
Other: sham acupuncture — different body acupuncture points will be selected to be manually punctured in addition to 4 acupoints on the skin of abdominal surface (the four points will be electrical stimulated during acupuncture). opposite to group A, in this group, the acupuncture needles will be inserted manually and very adjacent to the real location of group-A acupoints (sham acupuncture). The electrical stimulator will connected to abdominal acupoints (bilateral Stomach 25 in addition to gallbladder 28 acupoints) but it will be turned off during the sessions. the session will repeated thrice weekly. the total duration of the study will be 60 days
  Arms: Group B

SUMMARY:
nowadays, published literature affirms strong relation between tinnitus, obesity, and high lipids of blood.

DETAILED DESCRIPTION:
For 8 weeks, our study will search effect of acupuncture on tinnitus (chronic subjective type), lipids and weight reduction in obese persons.

ELIGIBILITY:
Inclusion Criteria:

* obese patients
* tinnitus complaints (chronic subjective form)

Exclusion Criteria:

* diabetics
* cardiovascular and neurogenic manifestations

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
tinnitus handicap inventory | It will be measured after eight weeks of acupuncture
  quality of life measure

SECONDARY OUTCOMES:
cholesterol | It will be measured after eight weeks of acupuncture
  serum lipid
triglycerides | It will be measured after eight weeks of acupuncture
  serum lipid
high density lipoprotein | It will be measured after eight weeks of acupuncture
  serum lipid
low density lipoproetin | It will be measured after eight weeks of acupuncture
  serum lipid
body mass index | It will be measured after eight weeks of acupuncture
  anthropometry measure
waist circumference | It will be measured after eight weeks of acupuncture
  anthropometry measure
visual analogue scale | It will be measured after eight weeks of acupuncture
  as a measure for severity of ear tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt